CLINICAL TRIAL: NCT04273620
Title: Randomized Controlled Trial of Combined Optokinetic Stimulation and Cueing-based Reading Therapy to Treat Hemispatial Neglect Following Stroke (OKS-READ Study)
Brief Title: Combined Optokinetic Stimulation and Cueing-based Reading Therapy to Treat Hemispatial Neglect Following Stroke
Acronym: OKS-READ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Bjoern Machner, Principal Investigator, Consultant Neurologist, University of Luebeck
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ULuebeck
Record Dates: First submitted 2020-02-07; First posted 2020-02-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Spatial Neglect

STUDY DESIGN:
Intervention Model Description: This study will be a mono-centric, randomized, controlled, clinical trial. Using a crossover design with two arms, patients will either receive the intervention therapy first and then the control treatment or they will start in the control arm and then switch to the intervention.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Due to the implicit constraints of cognitive interventions (no placebo possible as opposed to drug studies), neither the patient himself nor the therapist of the study can be blinded to the patient's allocation arm. However, the assessment of the functional impairment will be performed by rehabilitation staff who are blind to the patient's allocation. Furthermore, the assessment of neglect severity by use of a computerized neuropsychological test battery is robust and objective and largely independent of the investigator who is administering the test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Control (IC) (Experimental): In the Intervention-Control (IC) arm, patients will first receive the intervention (OKS-READ) containing 15 individual therapy sessions within a maximum time period of 28 days. Afterwards they will receive the control therapy (again 15 sessions within max. 28 days).
  Interventions: Behavioral: Optokinetic stimulation and cueing-based reading therapy (OKS-READ); Behavioral: General neuropsychological treatment
- Control-Intervention (CI) (Active Comparator): In the Control-Intervention (CI) arm, patients will first receive the control therapy (15 sessions within max. 28 days), followed by the intervention phase (15 therapy sessions OKS-READ within a maximum time period of 28 days).
  Interventions: Behavioral: Optokinetic stimulation and cueing-based reading therapy (OKS-READ); Behavioral: General neuropsychological treatment

INTERVENTIONS:
Behavioral: Optokinetic stimulation and cueing-based reading therapy (OKS-READ) — Each intervention session starts with an optokinetic stimulation (OKS) of at least 15 minutes duration. A pattern of squares, dots, triangles and stars will coherently and continuously move to the left on a computer screen in front of the patients. Patients are instructed to choose one stimulus and follow it with the eyes until it has reached the left side of the screen, then jump to the right edge of the screen and start again.
  The second part of each intervention session is the cueing-based reading therapy (READ), which will also last at least 15 minutes. The task of the patient is to read out loud words or a text presented on a paper in front of them. We will use exogenous (e.g., the therapist highlights words when they were omitted) and endogenous cues (verbal instructions which require intrinsic action by the patient) to facilitate attentional shifts to the left. The intensity of cueing will be matched to the actual severity of neglect (adaptive therapy).
Behavioral: General neuropsychological treatment — As a control treatment the patients will receive neuropsychological treatment without targeting visuospatial attention. Examples for components implemented are supporting conversations, diagnostic assessments (e.g. memory diagnostics) and training of memory and executive functions.

SUMMARY:
Spatial neglect represents a common and severe cognitive disorder following unilateral (mostly right hemisphere) stroke. Patients are unaware of objects, persons and even own body parts in the (usually left) hemispace opposite to their brain lesion. While there is spontaneous remission in some patients, neglect symptoms persist in many stroke survivors which is associated with a poor functional outcome. Although different therapeutic approaches (including cognitive interventions, non-invasive brain stimulation and drugs) have been investigated in the last decades, an established therapy is still missing. Hence, there is a clear need for an effective and feasible intervention that can be applied in rehabilitation centers.

This study is dedicated to assess the effect of a cognitive treatment consisting of combined optokinetic stimulation (OKS) and cueing-based reading therapy (READ) on hemispatial neglect and the neglect-related functional disability in right-hemisphere stroke patients. It will be a mono-centric, randomized, controlled, clinical trial. Using a crossover design with two arms, patients will either receive the intervention therapy (OKS-READ) first and subsequently the control treatment (neuropsychological training not targeting visuospatial attention) or they will start in the control arm and then switch to the intervention. Each treatment phase consists of 15 therapy sessions lasting 30 to 45 minutes. The outcome will be assessed at different time points, including established neuropsychological tests for spatial neglect and a clinical score of neglect-related functional disability.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* a first-time stroke in the right hemisphere (confirmed by cranial CT or MRI) within the last six months,
* a left-sided hemispatial neglect (as detected in at least one subtest of the neuropsychological test battery at screening),
* the ability to read and understand German language and
* the ability to give informed consent.

Exclusion Criteria:

* dementia
* other structural brain lesions besides the unilateral stroke (e.g. multiple or bilateral stroke lesions, hydrocephalus, inflammatory lesions, etc.)
* low vision (corrected <0.7) due to ophthalmological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Neglect symptom severity (neuropsychological test performance) | Intra-individual difference of the outcome's change during 3 weeks Intervention versus 3 weeks Control phase, i.e. (T3 on Day 21 - T2 on Day 1) - (T5 on Day 42 - T4 on Day 22)
  Composite score of different established computerized tests assessing spatial neglect (minimum 0%, maximum 100%, higher score means better outcome)
Neglect-related functional disability | Intra-individual difference of the outcome's change during 3 weeks Intervention versus 3 weeks Control phase, i.e. (T3 on Day 21 - T2 on Day 1) - (T5 on Day 42 - T4 on Day 22)
  Clinical score of neglect-related functional disability (Catherine Bergego Scale, CBS; minimum 0, maximum 30, higher score means worse outcome)

SECONDARY OUTCOMES:
Neglect dyslexia | Intra-individual difference of the outcome's change during 3 weeks Intervention versus 3 weeks Control phase, i.e. (T3 on Day 21 - T2 on Day 1) - (T5 on Day 42 - T4 on Day 22)
  Performance in the Menu reading task of the Behavioural Inattention Test battery (minimum 0 correct words (worst outcome), maximum 24 correct words (best outcome)
Attention bias during a visuo-motor cancellation task | Intra-individual difference of the outcome's change during 3 weeks Intervention versus 3 weeks Control phase, i.e. (T3 on Day 21 - T2 on Day 1) - (T5 on Day 42 - T4 on Day 22)
  Bias of the Center of Cancellation (CoC) during the Bells test (values between -1 (strongest leftward bias), 0 (no bias) and +1 (strongest rightward bias)
Oculomotor bias during visual exploration | Intra-individual difference of the outcome's change during 3 weeks Intervention versus 3 weeks Control phase, i.e. (T3 on Day 21 - T2 on Day 1) - (T5 on Day 42 - T4 on Day 22)
  Bias of the Center of Fixation (CoF) during free viewing of naturalistic photographs as measured with an infrared remote eye tracker (values between -1 (strongest leftward bias), 0 (no bias) and +1 (strongest rightward bias)
Anosognosia | Intra-individual difference of the outcome's change during 3 weeks Intervention versus 3 weeks Control phase, i.e. (T3 on Day 21 - T2 on Day 1) - (T5 on Day 42 - T4 on Day 22)
  Difference between investigator-assessed CBS score and the patient's self-assessed CBS score
Non-neglect specific functional outcome (Barthel) | Intra-individual difference of the outcome's change during 3 weeks Intervention versus 3 weeks Control phase, i.e. (T3 on Day 21 - T2 on Day 1) - (T5 on Day 42 - T4 on Day 22)
  Barthel Index (min. 0, max. 100, higher score means better outcome)
Functional Independence (FIM) | Intra-individual difference of the outcome's change during 3 weeks Intervention versus 3 weeks Control phase, i.e. (T3 on Day 21 - T2 on Day 1) - (T5 on Day 42 - T4 on Day 22)
  Functional Independence Measure (18 items scale with scores between 0 and 7 points; higher scores mean better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Bjoern Machner, MD, Principal Investigator — University of Luebeck
Locations (1):
- University of Luebeck, Dept. of Neurology, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bode LKG, Sprenger A, Helmchen C, Hauptmann B, Munte TF, Machner B. Combined optokinetic stimulation and cueing-assisted reading therapy to treat hemispatial neglect: A randomized controlled crossover trial. Ann Phys Rehabil Med. 2023 Jun;66(5):101713. doi: 10.1016/j.rehab.2022.101713. Epub 2023 Jan 14. PMID 36645965
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT04273620/Prot_SAP_000.pdf